CLINICAL TRIAL: NCT00001969
Title: Factors in Susceptibility to Ischemic Heart Disease in Major Depression: Documentation of Insulin Resistance in Patients With Major Depression Utilizing the Hyperinsulinemic Euglycemic Glucose Clamp
Brief Title: Heart Disease Risk Factors in Major Depression
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000049; 00-M-0049
Record Dates: First submitted 2000-01-18; First posted 2000-01-19 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-01-19

CONDITIONS: Adrenal Gland Hyperfunction; Cardiovascular Disease; Involutional Depression
Keywords: Cardiovascular Disease; Glucose Clamp; Hypercortisolism; Insulin Sensitivity; Major Depression Disorder; Inflammation; Coagulation; Metabolic; Insulin; Cytokine; Depression; Volunteer; Healthy Volunteer
MeSH Terms: conditions — Adrenocortical Hyperfunction; Cardiovascular Diseases; Depressive Disorder, Major; Cushing Syndrome; Insulin Resistance; Inflammation; Thrombosis; Depression

SUMMARY:
A series of studies in patients with major depression have consistently demonstrated a doubling of the mortality rate at any age, independent of suicide. In addition, the relative risk for clinically significant coronary artery disease in patients with major depression is also 2 or more in studies that independently controlled for risk factors such as smoking, hypertension, etc. The principal long-term goals of the CNE include the determination of the mechanisms that underlie enhanced susceptibility to premature ischemic heart disease in patients with major depression, documenting the age at which demonstrable pathophysiologic or predictive changes begin to occur, and charting their rate of progression. Our long-term goal is to use our understanding of underlying mechanisms to enhance our capacity to predict who with major depression is most likely to develop premature ischemic heart disease, to determine what the mechanisms underlying this susceptibility are, and to develop improved means for treatment and prevention.

Depressed patients are known to manifest a variety of neuroendocrine changes that predispose to coronary artery disease including hypercortisolism, decreased secretion of growth hormone and a deficiency of sex steroids. A final common denominator of these neuroendocrine abnormalities is insulin resistance. Insulin resistance promotes several changes that would favor hypertension and increased coronary artery disease including increased sodium retention, increased activity of the sympathetic nervous system, proliferation of vascular smooth muscle and deposition of highly metabolically active visceral fat. The latter induces additional risk factors for coronary disease, including dyslipidemia, hypercoagulation, and enhanced inflammation. It is a matter of public health importance to document the frequency and severity of insulin resistance in patients with major depression compared to a closely matched group of healthy controls. To accurately quantify insulin resistance in each patient and control, we will apply the hyperinsulinemic euglycemic glucose clamp procedure. This is the gold standard method for measuring the insulin sensitivity since it reflects the direct human body glucose metabolic response to a known insulin infusion. Moreover, it is essential to use this technique in patients with major depression as data indicate that other alternative procedures give unreliable results in the context of hypercortisolism.

DETAILED DESCRIPTION:
A series of studies in patients with major depression have consistently demonstrated a doubling of the mortality rate at any age, independent of suicide. In addition, the relative risk for clinically significant coronary artery disease in patients with major depression is also 2 or more in studies that independently controlled for risk factors such as smoking, hypertension, etc. The principal long-term goals of the CNE include the determination of the mechanisms that underlie enhanced susceptibility to premature ischemic heart disease in patients with major depression, documenting the age at which demonstrable pathophysiologic or predictive changes begin to occur, and charting their rate of progression. Our long-term goal is to use our understanding of underlying mechanisms to enhance our capacity to predict who with major depression is most likely to develop premature ischemic heart disease, to determine what the mechanisms underlying this susceptibility are, and to develop improved means for treatment and prevention.

Depressed patients are known to manifest a variety of neuroendocrine changes that predispose to coronary artery disease including hypercortisolism, decreased secretion of growth hormone and a deficiency of sex steroids. A final common denominator of these neuroendocrine abnormalities is insulin resistance. Insulin resistance promotes several changes that would favor hypertension and increased coronary artery disease including increased sodium retention, increased activity of the sympathetic nervous system, proliferation of vascular smooth muscle and deposition of highly metabolically active visceral fat. The latter induces additional risk factors for coronary disease, including dyslipidemia, hypercoagulation, and enhanced inflammation. It is a matter of public health importance to document the frequency and severity of insulin resistance in patients with major depression compared to a closely matched group of healthy controls. To accurately quantify insulin resistance in each patient and control, we will apply the hyperinsulinemic euglycemic glucose clamp procedure. This is the gold standard method for measuring the insulin sensitivity since it reflects the direct human body glucose metabolic response to a known insulin infusion. Moreover, it is essential to use this technique in patients with major depression as data indicate that other alternative procedures give unreliable results in the context of hypercortisolism.

ELIGIBILITY:
* INCLUSION CRITERIA

Adults between the ages of 21 and 55, with or without major depression as diagnosed with The Structured Clinical Interview of Diagnosis (SCID) of the Diagnostic and Statistical Manual of Mental Disorder, Fourth Edition (DSM-IV), will be recruited. All depressed patients will be included, although we will characterize patients a priori as having a predominantly melancholic, atypical, or mixed symptom pattern. We plan to recruit at least 20 patients in each group.

Both currently depressed patients (greater than 14 on the Hamilton Depression Rating Scale) and those with a history of major depression who are clinically recovered will be included. Patients may be taking psychotropic medications for depression at the time of study. Sub-analyses will be done comparing steady-state glucose utilization rates as a function of mood state and medication status. Subjects should not have significant underlying illnesses known to affect insulin sensitivity, and should have a body mass index between 20 and 30 kg/m2.

EXCLUSION CRITERIA

1. Pregnancy
2. Existing diabetes mellitus
3. Body mass index less than 20 or greater than 30 kg/ m2
4. Existing cardiovascular diseases and other end organ diseases
5. Existing peripheral vascular disease
6. HIV infection
7. Patients who are on B-blockers, thiazides, and/or glucocorticoids and cannot discontinue these medications.
8. Subjects who are on oral contraceptives need to discontinue the medication for 1-2 days before the clamp study.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160
Dates: Start 1999-12-30; Study Completion 2007-01-19

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Anda RF, Williamson DF, Escobedo LG, Mast EE, Giovino GA, Remington PL. Depression and the dynamics of smoking. A national perspective. JAMA. 1990 Sep 26;264(12):1541-5. PMID 2395193